CLINICAL TRIAL: NCT06831045
Title: A Clinical Comparison in Wound Healing of Bikini Versus Longitudinal Incision in Direct Anterior Approach Total Hip Arthroplasty in the Obese Patient Population: A Randomized Control Trial
Brief Title: Bikini vs Longitudinal Incision in Direct Anterior Approach (DAA) Total Hip Arthroplasty (THA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor of Clinical Orthopedics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230334
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: THA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bikini Incision Group (Experimental): Participants in this group will receive the bikini incision during THA. Total participation is up to 90 days.
  Interventions: Procedure: Bikini Incision
- Longitudinal Incision Group (Experimental): Participants in this group will receive the longitudinal incision during THA. Total participation is up to 90 days.
  Interventions: Procedure: Longitudinal Incision

INTERVENTIONS:
Procedure: Bikini Incision — Participants will receive the bikini incision in person during THA. A one-time incision will be made along the groin line before standard of care THA surgery. The surgery takes approximately two hours.
  Arms: Bikini Incision Group
Procedure: Longitudinal Incision — Participants will receive the longitudinal incision in person during THA. A one-time linear incision will be made along the thigh before standard-of-care THA surgery. The surgery takes approximately two hours.
  Arms: Longitudinal Incision Group

SUMMARY:
The study team is conducting this study to see if there is a difference between the wound healing and participant satisfaction rates between two incision types used during a THA done via the DAA technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index greater than or equal to 30
* Patients undergoing primary unilateral DAA THA
* Patients undergoing primary THA

Exclusion Criteria:

* Patients with body mass index less than 30
* Patients with a history of prior open surgery on the affected hip
* Patients unable/unwilling to undergo spinal anesthesia under monitored anesthesia care (MAC)
* Patients with allergies or absolute contraindication to standardized drugs administered within the University of Miami protocol for total hip replacement
* The following groups will not be included: adults unable to consent, individuals who are not yet adults, pregnant women, prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Wound Healing measured in number of days | Up to 14 days
  Will be measured in number of days the incision will take to heal.
Patient satisfaction with scaring as measured by Patient Scar Assessment Scale | Up to to 6 months
  Score ranges from 0 to 10. Higher scores indicate less satisfaction
Scar cosmesis as measured by Observer Scar Assessment Scale | Up to 6 months
  Score ranges from 0 to 10. Higher scores indicate worse scar cosmesis

SECONDARY OUTCOMES:
Number of participants who report lateral femoral cutaneous nerve-related symptoms | Up to 6 months
  Number of participants who report lateral femoral cutaneous nerve-related symptoms
Patient reported outcomes as measured by Hip Disability and Osteoarthritis Outcomes | Up to 6 months
  Scores range from 0 to 28. Higher scores indicate worse patient reported outcomes
Number of intraoperative fractures | Up to 3 hours
  Number of intraoperative fractures
Length of surgery measured in minutes | Up to 3 hours
  Length of surgery measured in minutes
Number of postoperative complications | Up to 90 days
  Number of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No